CLINICAL TRIAL: NCT00294489
Title: Methacetin Breath Test in HCV Patients With Normal and Near-Normal ALT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: ORHCV1-HMO-CTIL
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2006-02

CONDITIONS: Chronic Hepatitis C Virus Infection
Keywords: HCV; Fibrosis; Breath test
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
A relatively large proportion of patients with chronic HCV infection have normal or mildly elevated ALT. Many of these patients are not being treated, and are not being sent for a liver biopsy. The present study will determine the ability of Methcetin BreathID Test(MBIT) to detect those patients who will be candidates for anti-viral treatment, as an alternative measure for liver biopsy in decision-making prior to treatment in clinical hepatology.

DETAILED DESCRIPTION:
The rational for using MBIT in the management of HCV in patients with persistently normal (and slightly elevated) ALT:

* If MBIT is impaired, this indicates fibrosis >2: a trigger to begin treatment
* This strategy will enable treating patients with relatively severe disease that was not detected by biopsy.
* HMOs recognize the cost-effectiveness of anti-viral therapy in these patients, as a means of prevention of deterioration, cirrhosis and HCC.
* If MBIT indicates low fibrosis => treatment may be deferred, and follow-up is performed to detect any possible degradation that will indicate need for treatment.
* Today the AASLD guidelines allow for treatment of HCV RNA+ patients with normal ALT. In view of the limited effectivity of therapy, its cost and side effects, there are likely to be many individuals in whom therapy can be safely deferred, leading to cost saving.
* MBIT may replace the need of liver biopsy for decision- making in HCV.
* Even in patients with genotype 1 and elevated ALT, or with risk of side effects, treatment may be delayed in low fibrosis (e.g. <2).

GOAL:

• To assess the ability of the MBIT to improve the management of patients for liver disorders

AIM:

• To determine whether the Methacetin BreathID Test (MBIT) can be useful in evaluation of HCV RNA positive patients with normal or minimally elevated ALT and to determine the severity of their liver disease as a guide for decision-making in routine clinical use.

OBJECTIVE:

AUC>0.75 (+/-10% in 95%CI) in detection of fibrosis>2.

INCLUSION CRITERIA:

* Men or women>18
* Patients with HCV RNA+ above 105 copies Patients with normal liver enzymes on two tests 3 months apart, or up to <X1.5 of upper normal
* Patients with biopsy proven HCV or (9 months prior to test with no anticipated changes in liver disease since biopsy).

EXCLUSION CRITERIA:

* Other liver disorders.
* Active infections.
* Use of drugs that are known to induce/suppress P4501A2
* Pulmonary diseases
* Consumption of >20cc alcohol a day prior to the test.

NUMBER OF PATIENTS:

* 200 HCV
* 50 matched controls

METHODS:

* Patient selection - All the patients that underwent a liver biopsy in the last 9 months in each center are invited to participate in the study, assuming they meet inclusion/exclusion criteria.
* Patients will undergo MBIT and data will be compared with the results of the different fibrotic and inflammatory scores (i.e. METAVIR) on liver biopsy. One pathologist will re-examine all biopsies.
* Oridion BreathID will provide MBIT data on 50 healthy controls.
* Substrate - A test meal consisting of 75mg PO methacetin + a known surface-active ingredient routinely used in the food and drug industry.
* Test length - 1 hour
* Fasting-8 hours fast only.
* The patient will be attached to the BreathID device via a nasal cannula and after baseline breath is measured, the test meal will be ingested and the device will continue measuring the exhaled breath for 1 hour. The BreathID device automatically measures changes in the 13C/12C ratio due to metabolization of the methacetin, using a spectroscopic principal. The results are printed out automatically at the end of the test.

STUDY DESIGN:

• At first visit to physician, patients will perform viral load test, liver enzymes tests and MBIT. A biopsy will have been performed within 9 months of these tests.

ELIGIBILITY:
Inclusion Criteria:

* Men or women>18
* Patients with HCV RNA+ above 105 copies Patients with normal liver enzymes on two tests 3 months apart, or up to <X1.5 of upper normal
* Patients with biopsy proven HCV or (9 months prior to test with no anticipated changes in liver disease since biopsy).

Exclusion Criteria:

* Other liver disorders.
* Active infections.
* Use of drugs that are known to induce/suppress P4501A2
* Pulmonary diseases
* Consumption of >20cc alcohol a day prior to the test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2006-02; Study Completion 2006-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gadi Lalazar, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Braden B, Faust D, Sarrazin U, Zeuzem S, Dietrich CF, Caspary WF, Sarrazin C. 13C-methacetin breath test as liver function test in patients with chronic hepatitis C virus infection. Aliment Pharmacol Ther. 2005 Jan 15;21(2):179-85. doi: 10.1111/j.1365-2036.2005.02317.x. PMID 15679768
- See also: Company producing Breath ID machine and substances — http://oridion.com